CLINICAL TRIAL: NCT01459172
Title: Human Breast Tissue Bioavailability of Topically Applied Limonene
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 07-0375-04
Record Dates: First submitted 2011-10-20; First posted 2011-10-25 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2011-10

CONDITIONS: Breast Cancer
Keywords: breast cancer prevention
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Limonene intervention (Experimental)
  Interventions: Other: limonene containing massage oil

INTERVENTIONS:
Other: limonene containing massage oil — daily massage application to the breast for 4 weeks

SUMMARY:
The overall objective of this project is to determine the safety and breast tissue bioavailability of limonene following massage application of limonene containing massage oil to the breast.

ELIGIBILITY:
Inclusion Criteria:

* Women who are 18-65 years of age
* ECOG performance status 0-1
* Normal organ and marrow function
* Women of child-bearing potential must agree to use adequate contraception
* Willing to avoid consumption and use of citrus or citrus containing products throughout the study
* Have both breasts intact

Exclusion Criteria:

* Have had cancer(s) within the past 5 years
* Participated in another clinical interventional trial within the past 3 months
* Uncontrolled intercurrent illness
* Pregnant or breast feeding
* Unable to produce nipple aspirate fluid
* Have known allergic or sensitive reactions to skin care products, citrus or coconut oil
* Have ongoing skin disorders such as eczema and psoriasis

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2007-10; Primary Completion 2010-02 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
breast tissue bioavailability | 4 weeks
  limonene levels in nipple aspirate fluid after 4 weeks of intervention

SECONDARY OUTCOMES:
safety | 6 weeks
  number of participants with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Sherry Chow, Ph.D., Principal Investigator — The University of Arizona
Locations (1):
- The University of Arizona Cancer Center, Tucson, Arizona, United States